CLINICAL TRIAL: NCT02422745
Title: COcoa Supplement and Multivitamin Outcomes Study
Acronym: COSMOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); Mars, Inc. (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, JoAnn E. Manson, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2014P002768
Record Dates: First submitted 2015-04-17; First posted 2015-04-21 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Disease; Cancer
Keywords: Cocoa extract multivitamins cardiovascular disease cancer
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms | interventions — Chocolate; Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cocoa extract + multivitamin (Active Comparator)
  Interventions: Dietary Supplement: Cocoa extract; Dietary Supplement: Multivitamin
- Cocoa extract + multivitamin placebo (Active Comparator)
  Interventions: Dietary Supplement: Cocoa extract; Dietary Supplement: Multivitamin placebo
- Cocoa extract placebo + multivitamin (Active Comparator)
  Interventions: Dietary Supplement: Multivitamin; Dietary Supplement: Cocoa extract placebo
- Cocoa extract placebo + multivitamin placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Cocoa extract placebo; Dietary Supplement: Multivitamin placebo

INTERVENTIONS:
Dietary Supplement: Cocoa extract — 2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin, and 50 mg theobromine
  Arms: Cocoa extract + multivitamin; Cocoa extract + multivitamin placebo
Dietary Supplement: Multivitamin — Multivitamin
  Arms: Cocoa extract + multivitamin; Cocoa extract placebo + multivitamin
Dietary Supplement: Cocoa extract placebo — Cocoa extract placebo
  Arms: Cocoa extract placebo + multivitamin; Cocoa extract placebo + multivitamin placebo
Dietary Supplement: Multivitamin placebo — Multivitamin placebo
  Arms: Cocoa extract + multivitamin placebo; Cocoa extract placebo + multivitamin placebo

SUMMARY:
The purpose of this study is to determine whether taking daily, dietary supplements of cocoa extract (containing cocoa flavanols and theobromine from the cocoa bean) and/or a standard multivitamin reduces the risk of developing cardiovascular disease (including heart attack, stroke, coronary revascularization, unstable angina or acute coronary syndrome (ACS) requiring hospitalization, carotid artery surgery, and peripheral artery surgery or angioplasty, and cardiovascular mortality) and cancer.

DETAILED DESCRIPTION:
The COcoa Supplement and Multivitamin Outcomes Study (COSMOS) is a randomized clinical trial of cocoa extract supplement (containing a total of 600 mg/d cocoa flavanols, including 80 mg. (-)-epicatechins), and a standard multivitamin supplement to reduce the risk of cardiovascular disease and cancer among women aged 65 years and older and men aged 60 years and older.

After the COSMOS trial began, an advanced method to analyze cocoa flavanols was accredited by AOAC International as a First Action Official Method of Analysis (https://doi.org/10.1093/jaoacint/qsaa132). This updated method relies on a reference material (RM8403) recently standardized and made commercially available by the U.S. National Institute of Standards and Technology. While the actual cocoa flavanol content of the COSMOS intervention remained unchanged throughout the trial, the application of this new analytical method led to expected changes in how the total cocoa flavanol content is now reported. Applying AOAC 2020.05/RM8403 to the COSMOS intervention, the total cocoa flavanol content of the COSMOS intervention is now 500 mg/day. Reporting of (-)-epicatechin content remained unaffected. Going forward, we will therefore apply AOAC 2020.05/RM8403 and report that the COSMOS intervention tested 500 mg/day of cocoa flavanols, including 80 mg of (-)-epicatechin.

Participants in COSMOS were recruited from among Women's Health Initiative (WHI) Extension Study cohort members; non-randomized respondents to mailings for the VITamin D and OmegA-3 TriaL (VITAL); respondents to nationwide invitational mailings to age-eligible adults; and volunteers who learned about the trial through the media or through ResearchMatch.org, an electronic recruitment website.

Several small randomized trials have demonstrated benefits for cocoa flavanols on intermediate outcomes, including blood pressure, lipids, insulin sensitivity, and flow-mediated vasodilation. For multivitamins, a prior large-scale randomized trial in middle-aged and older men showed a significant reduction in cancer, but comparable trial data in women are lacking. For both interventions, a large-scale clinical trial such as COSMOS could have major clinical and public health implications.

Eligible participants have been assigned by chance (like a coin toss) to one of four groups: (1) daily cocoa extract and multivitamin; (2) daily cocoa extract and multivitamin placebo; (3) daily cocoa extract placebo and multivitamin; or (4) daily cocoa extract placebo and multivitamin placebo. Participants have an equal chance of being assigned to any of these four groups and a 3 out of 4 chance of receiving at least one active agent.

Participants in all groups take three pills each day: two capsules that contain either cocoa extract or cocoa extract placebo, and one tablet that contains either multivitamin or multivitamin placebo. Participants receive their study pills in convenient calendar packs via U.S. mail.

Participants are asked to complete mailed questionnaires each year. The questionnaires ask about health; lifestyle habits, such as diet, physical activity, and smoking; use of medications and dietary supplements; family history of illness and new medical diagnoses. Occasionally, participants may receive a phone call from study staff to collect information or clarify responses on the questionnaires.

The expected rates for our original primary composite cardiovascular disease (CVD) endpoint were based on the projected age and sex distribution of the trial cohort and CVD event rates from our previously conducted trials. However, we determined that the observed rates of CVD endpoints among COSMOS participants were lower than expected due to a younger population of women, increasing use of statins and other pharmacotherapies as seen in other recently published clinical trials, and the impact of COVID-19 on fewer reports of CVD diagnoses, hospitalizations, and procedures. As a result, the COSMOS Data and Safety Monitoring Board (DSMB) approved a proposal to add three new outcomes to our primary composite CVD endpoint: (1) unstable angina or acute coronary syndrome requiring hospitalization, (2) carotid artery surgery, and (3) peripheral artery surgery or angioplasty. These additional CVD outcomes are consistent with the atherosclerotic mechanisms underlying the postulated effects for the randomized interventions. COSMOS participants have already provided self-reports of these diagnoses since the start of the COSMOS trial that will be adjudicated via medical records. The original primary composite CVD endpoint will still be evaluated as a secondary outcome.

At baseline, approximately 7,000 COSMOS participants provided optional blood and urine samples, which will be used to determine whether the study agents significantly change biomarkers and other risk factors related to cardiovascular disease and cancer. Selected participants either have specimens collected through mailed specimen collection kits that are returned by the participant, or have blood, urine, blood pressure, and anthropometric measurements collected by technicians from Examination Management Services, Inc. (EMSI), a national clinical services provider. A subgroup of those who provide baseline specimens and measurements are asked to provide follow-up samples and measurements.

At baseline and year 2 of the trial, approximately 600 participants living within driving distance of Boston, Massachusetts provide additional measurements from in-clinic study visits at the Clinical and Translational Science Center (CTSC) of Brigham and Women's Hospital. These visits include cognitive function assessments, anthropometrics, physical function assessments, blood pressure and other measurements. The trial will assess whether the study agents significantly affect changes in these variables over time.

Primary Hypotheses:

1. A cocoa extract supplement will reduce the risk of major cardiovascular events, defined as a composite endpoint of myocardial infarction, stroke, cardiovascular mortality, coronary revascularization, unstable angina or ACS requiring hospitalization, carotid artery surgery, and peripheral artery surgery or angioplasty;
2. A daily multivitamin will reduce the risk of invasive cancer (excluding non-melanoma skin cancer).

Secondary Hypotheses:

1. Cocoa extract will reduce the risk of a composite endpoint of MI, stroke, cardiovascular mortality, and coronary revascularization;
2. Cocoa extract will reduce the risk of invasive cancer (excluding non-melanoma skin cancer);
3. A daily multivitamin will reduce the risk of major cardiovascular events;
4. Cocoa extract and/or a daily multivitamin will reduce the combined endpoint of major cardiovascular events plus all-cause mortality;
5. Cocoa extract and/or a daily multivitamin will reduce the risk of individual cardiovascular events, including myocardial infarction, stroke, cardiovascular mortality, coronary revascularization, unstable angina or ACS requiring hospitalization, carotid artery surgery, and peripheral artery surgery or angioplasty, and total mortality; plus site-specific cancers, including breast, colorectal, and lung cancer;
6. A daily multivitamin will reduce the risk of cancer among women and men with a history of cancer at baseline;
7. In a subset of equal numbers of female and male COSMOS respondents who provide baseline bloods and/or urine samples, cocoa extract and/or a daily multivitamin will significantly change blood and/or urinary levels of flavonoids or their metabolites from baseline to 1, 2, or 3 years of follow-up.

Tertiary Aim:

To assess whether the cocoa extract and/or a daily multivitamin exhibit synergistic effects on risk of major cardiovascular events or cancer, and if the effects vary by nutritional status or medication use.

Aims of Clinical and Translational Science Center (CTSC) Component:

To test whether the cocoa extract and/or a daily multivitamin has beneficial effects on:

1. Systolic and diastolic blood pressure;
2. Pulse wave velocity (PWV) and central blood pressure indices as measured by pulse wave analysis;
3. Cognitive function and memory;
4. Physical performance as assessed by balance tests, grip strength, timed chair stands, and walking speed,
5. Bone loss in the spine, hip and total body as assessed by bone-mineral density (BMD) and changes in body composition as assessed by dual x-ray absorpiometry (DXA);

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 65 years of age participating in the Women's Health Initiative (WHI) Extension Study.
2. Men ≥ 60 years of age and women age ≥ 65 years of age who were contacted for but not randomized into the VITAL trial.
3. Other women ≥ 65 years of age and men aged ≥ 60 years of age who responded to targeted mass mailings and volunteers who learned about the trial through the media or through ResearchMatch.org, an electronic recruitment website.
4. Willing to participate, as evidenced by providing informed consent and completing all required baseline forms.

Exclusion Criteria:

1. History of myocardial infarction or stroke.
2. Diagnosed with invasive cancer other than non-melanoma skin cancer in the last 2 years prior to enrollment.
3. Any serious illness that would preclude participation and/or completion of the trial, including the diagnosis of kidney failure and current dialysis treatment.
4. Taking cocoa extract or multivitamin supplements and not willing to forego use during the trial.
5. Taking total supplemental vitamin D > 1,000 IU/day and not willing to forego use during the trial.
6. Taking total supplemental calcium > 1,200 mg/day and not willing to forego use during the trial.
7. Extreme sensitivity to caffeine.
8. Consume < 75% of the expected number of both types of supplements during the run-in phase.
9. Unable to communicate in English due to language barrier or mental incapacity.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21442 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn E. Manson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Hamaya R, Li S, Lau J, Rautiainen S, Haring B, Liu S, Shadyab AH, Martin LW, Wassertheil-Smoller S, Rist PM, Manson JE, Sesso HD; COSMOS Research Group. Long-term effect of multivitamin supplementation on incident self-reported hypertension and blood pressure changes in the COSMOS trial. Am J Hypertens. 2025 Nov 20:hpaf224. doi: 10.1093/ajh/hpaf224. Online ahead of print. PMID 41264477
- [Derived] Vyas CM, Manson JE, Sesso HD, Cook NR, Rist PM, Weinberg A, Moorthy MV, Baker LD, Espeland MA, Yeung LK, Brickman AM, Okereke OI. Effect of multivitamin-mineral supplementation versus placebo on cognitive function: results from the clinic subcohort of the COcoa Supplement and Multivitamin Outcomes Study (COSMOS) randomized clinical trial and meta-analysis of 3 cognitive studies within COSMOS. Am J Clin Nutr. 2024 Mar;119(3):692-701. doi: 10.1016/j.ajcnut.2023.12.011. Epub 2024 Jan 18. PMID 38244989
- [Derived] Vyas CM, Manson JE, Sesso HD, Rist PM, Weinberg A, Kim E, Moorthy MV, Cook NR, Okereke OI. Effect of cocoa extract supplementation on cognitive function: results from the clinic subcohort of the COSMOS trial. Am J Clin Nutr. 2024 Jan;119(1):39-48. doi: 10.1016/j.ajcnut.2023.10.031. Epub 2023 Dec 7. PMID 38070683
- [Derived] Sesso HD, Rist PM, Aragaki AK, Rautiainen S, Johnson LG, Friedenberg G, Copeland T, Clar A, Mora S, Moorthy MV, Sarkissian A, Wactawski-Wende J, Tinker LF, Carrick WR, Anderson GL, Manson JE; COSMOS Research Group. Multivitamins in the prevention of cancer and cardiovascular disease: the COcoa Supplement and Multivitamin Outcomes Study (COSMOS) randomized clinical trial. Am J Clin Nutr. 2022 Jun 7;115(6):1501-1510. doi: 10.1093/ajcn/nqac056. PMID 35294969
- [Derived] Sesso HD, Manson JE, Aragaki AK, Rist PM, Johnson LG, Friedenberg G, Copeland T, Clar A, Mora S, Moorthy MV, Sarkissian A, Carrick WR, Anderson GL; COSMOS Research Group. Effect of cocoa flavanol supplementation for the prevention of cardiovascular disease events: the COcoa Supplement and Multivitamin Outcomes Study (COSMOS) randomized clinical trial. Am J Clin Nutr. 2022 Jun 7;115(6):1490-1500. doi: 10.1093/ajcn/nqac055. PMID 35294962
- [Derived] Rist PM, Sesso HD, Johnson LG, Aragaki AK, Wang L, Rautiainen S, Hazra A, Tobias DK, LeBoff MS, Schroeter H, Friedenberg G, Copeland T, Clar A, Tinker LF, Hunt RP, Bassuk SS, Sarkissian A, Smith DC, Pereira E, Carrick WR, Wion ES, Schoenberg J, Anderson GL, Manson JE; COSMOS Research Group. Design and baseline characteristics of participants in the COcoa Supplement and Multivitamin Outcomes Study (COSMOS). Contemp Clin Trials. 2022 May;116:106728. doi: 10.1016/j.cct.2022.106728. Epub 2022 Mar 12. PMID 35288332
- [Derived] Baker LD, Rapp SR, Shumaker SA, Manson JE, Sesso HD, Gaussoin SA, Harris D, Caudle B, Pleasants D, Espeland MA; COSMOS-Mind Research Group. Design and baseline characteristics of the cocoa supplement and multivitamin outcomes study for the Mind: COSMOS-Mind. Contemp Clin Trials. 2019 Aug;83:57-63. doi: 10.1016/j.cct.2019.06.019. Epub 2019 Jul 2. PMID 31271875
- See also: COSMOS Trial website — https://www.cosmostrial.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 191769 initially screened; 35669 eligible to enter run-in; 21442 eligible for randomization; 2x2 factorial design; 10719 assigned to active cocoa extract (of these, 5360 were assigned to active multivitamin and 5359 to placebo multivitamin) & 10723 assigned to placebo cocoa extract (of these, 5360 were assigned to active multivitamin and 5363 to placebo multivitamin)
Pre-assignment Details: The trial included at least a 2-month placebo run-in period to select participants likely to have excellent compliance. Only individuals who reported taking at least 75% or more of their their study pills during the run-in and met other eligibility criteria were randomized into the trial.
Groups:
- ACTIVE Cocoa Extract + ACTIVE Multivitamin: Cocoa extract: 2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin, and 50 mg theobromine
  Multivitamin: Multivitamin
- ACTIVE Cocoa Extract + PLACEBO Multivitamin: Cocoa extract: 2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin, and 50 mg theobromine
  Multivitamin placebo: Multivitamin placebo
- PLACEBO Cocoa Extract + ACTIVE Multivitamin: Multivitamin: Multivitamin
  Cocoa extract placebo: Cocoa extract placebo
- PLACEBO Cocoa Extract + PLACEBO Multivitamin: Cocoa extract placebo: Cocoa extract placebo
  Multivitamin placebo: Multivitamin placebo
Period: Overall Study
Arm/Group | ACTIVE Cocoa Extract + ACTIVE Multivitamin | ACTIVE Cocoa Extract + PLACEBO Multivitamin | PLACEBO Cocoa Extract + ACTIVE Multivitamin | PLACEBO Cocoa Extract + PLACEBO Multivitamin
Started | 5360 | 5359 | 5360 | 5363
Completed | 5360 | 5359 | 5360 | 5363
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ACTIVE Cocoa Extract + ACTIVE Multivitamin: Cocoa extract: 2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin and 50 mg theobromine
  Multivitamin: Multivitamin
- ACTIVE Cocoa Extract + PLACEBO Multivitamin: Cocoa extract: 2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin and 50 mg theobromine
  Multivitamin placebo: Multivitamin placebo
- Total: Total of all reporting groups
Arm/Group | ACTIVE Cocoa Extract + ACTIVE Multivitamin | ACTIVE Cocoa Extract + PLACEBO Multivitamin | PLACEBO Cocoa Extract + ACTIVE Multivitamin | PLACEBO Cocoa Extract + PLACEBO Multivitamin | Total
Number analyzed (Participants) | 5360 | 5359 | 5360 | 5363 | 21442
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 675 | 676 | 676 | 678 | 2705
  >=65 years | 4685 | 4683 | 4684 | 4685 | 18737
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (6.6) | 72.1 (6.6) | 72.1 (6.5) | 72.1 (6.5) | 72.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3171 | 3166 | 3167 | 3162 | 12666
  Male | 2189 | 2193 | 2193 | 2201 | 8776
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4796 | 4828 | 4832 | 4838 | 19294
  Black | 290 | 268 | 278 | 295 | 1131
  Asian/Pacific Islander | 138 | 136 | 120 | 105 | 499
  American Indian/Alaskan Native | 17 | 14 | 20 | 8 | 59
  Multiracial/other/unknown or not reported | 119 | 113 | 110 | 117 | 459
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 134 | 118 | 150 | 142 | 544
Region of Enrollment [Number; unit: participants]
  United States | 5360 | 5359 | 5360 | 5363 | 21442
Education [Count of Participants; unit: Participants]
  High school diploma/GED or less | 588 | 553 | 592 | 563 | 2296
  Attended or graduated from college | 2117 | 2211 | 2198 | 2159 | 8685
  Post-college | 2596 | 2551 | 2508 | 2586 | 10241
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.6 (5.3) | 27.7 (5.4) | 27.7 (5.4) | 27.8 (5.5) | 27.7 (5.4)
Cocoa extract use before run-in [Count of Participants; unit: Participants] — Participants had to agree to forgo cocoa extract supplements (chocolate intake was not restricted) during the trial.
  Participants | 22 | 23 | 20 | 26 | 91
Multivitamin use before run-in [Count of Participants; unit: Participants] — Participants had to agree to forgo multivitamin use during the trial.
  Participants | 2237 | 2201 | 2176 | 2181 | 8795
Chocolate intake [Count of Participants; unit: Participants] — Includes consumption of milk chocolate, dark chocolate, white chocolate and candy bars.
  Participants
    Rarely | 850 | 790 | 850 | 862 | 3352
    Monthly | 716 | 739 | 751 | 717 | 2923
    Weekly | 2800 | 2806 | 2775 | 2748 | 11129
    At least daily | 568 | 566 | 586 | 597 | 2317
History of cardiovascular disease [Count of Participants; unit: Participants] — This includes a history at baseline of coronary artery bypass graft (CABG)/percutaneous coronary intervention (PCI), unstable angina including hospitalization, carotid artery surgery/stenting, or peripheral artery surgery/stenting.
  Participants | 336 | 290 | 307 | 336 | 1269
Personal history of cancer [Count of Participants; unit: Participants] | 917 | 858 | 896 | 879 | 3550
History of diabetes [Count of Participants; unit: Participants] | 702 | 715 | 713 | 734 | 2864
History of hypertension [Count of Participants; unit: Participants] | 3048 | 3142 | 3105 | 3128 | 12423
Cholesterol-lowering medication use [Count of Participants; unit: Participants] | 2366 | 2346 | 2348 | 2345 | 9405
Aspirin use in past month [Count of Participants; unit: Participants] | 2617 | 2594 | 2551 | 2617 | 10379
Smoking status [Count of Participants; unit: Participants]
  Current | 199 | 199 | 218 | 219 | 835
  Past | 2173 | 2223 | 2172 | 2163 | 8731
  Never | 2904 | 2862 | 2904 | 2895 | 11565

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Total Cardiovascular Disease (CVD) Events
Description: CVD events include myocardial infarction, stroke, cardiovascular deaths, coronary revascularization procedures, unstable angina or acute coronary syndrome (ACS) requiring hospitalization, carotid artery surgery, and peripheral artery surgery or angioplasty. CVD events are confirmed by review of discharge summaries, ECG's, laboratory reports, test reports, radiology reports, surgical reports, medical records for reports of increased pain, use of medication to alleviate pain, and evidence of troponin leak, and death certificates.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Groups:
- Active Cocoa Extract: Cocoa extract: 2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin and 50 mg theobromine
- Cocoa Extract Placebo: Cocoa extract placebo, 2 capsules/day
- Active Multivitamin: Multivitamin, 1 tablet/day
- Multivitamin Placebo: Multivitamin placebo, 1 tablet/day
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 410 | 456 | 429 | 437

2. Primary Outcome: Number of Participants With Invasive Cancer Events
Description: Diagnoses of invasive cancer are confirmed by review of discharge summaries, pathology reports, operative reports, surgical reports, and diagnostic or treatment procedure reports, including both inpatient and outpatient procedures.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 550 | 503 | 518 | 535

3. Secondary Outcome: Number of Participants With Composite Endpoint of MI, Stroke, Cardiovascular Mortality, and Coronary Revascularization
Description: This outcome was a composite of myocardial infarction, stroke, cardiovascular deaths, and coronary revascularization procedures.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 362 | 403 | 381 | 384

4. Secondary Outcome: Number of Participants With Total Cardiovascular Events Plus All-Cause Mortality
Description: This outcome was a composite of myocardial infarction, stroke, cardiovascular deaths, coronary revascularization procedures, unstable angina or acute coronary syndrome (ACS) requiring hospitalization, carotid artery surgery, and peripheral artery surgery or angioplasty, plus all-cause mortality.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 665 | 731 | 680 | 716

5. Secondary Outcome: Number of Participants With Myocardial Infarction
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 88 | 101 | 96 | 93

6. Secondary Outcome: Number of Participants With Stroke
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 113 | 124 | 121 | 116

7. Secondary Outcome: Number of Participants With Cardiovascular Mortality
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 76 | 104 | 84 | 96

8. Secondary Outcome: Number of Participants With Coronary Revascularization
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 166 | 175 | 177 | 164

9. Secondary Outcome: Number of Participants With Unstable Angina or Acute Coronary Syndrome Requiring Hospitalization
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 46 | 46 | 50 | 42

10. Secondary Outcome: Number of Participants With Carotid Artery Surgery
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 25 | 27 | 24 | 28

11. Secondary Outcome: Number of Participants With Peripheral Artery Surgery or Angioplasty
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 17 | 19 | 16 | 20

12. Secondary Outcome: Number of Participants With Total Mortality
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 353 | 397 | 362 | 388

13. Secondary Outcome: Number of Participants With Breast Cancer
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 99 | 81 | 93 | 87

14. Secondary Outcome: Number of Participants With Colorectal Cancer
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 38 | 29 | 38 | 29

15. Secondary Outcome: Number of Participants With Lung Cancer
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 10719 | 10723 | 10720 | 10722
Participants | 49 | 58 | 41 | 66

16. Secondary Outcome: Median Urinary gVLM Levels at Year 2 Among Those Providing Spot Urine at Baseline and Year 2
Description: Baseline biospecimens were obtained during the run-in period from 6867 (32.0%) of 21,442 randomized participants, of whom 2050 participants comprised a longitudinal subcohort providing a baseline and at least one follow-up blood and/or spot urine sample at 1, 2, and/or 3 years follow-up. This includes 1,917 participants specifically providing spot urine samples at baseline and Year 2. From the spot urine samples collected, habitual flavanol consumption was estimated by urinary concentrations of 5-(3',4'-dihydroxyphenyl)-γ-valerolactone metabolite (gVLM), which are a biomarker of flavanol intake.
Time Frame: 2 years
Population: Within the subcohort providing a baseline and follow-up biospecimen, gVLM levels were analyzed from spot urine samples collected from 1,917 participants at 2 years follow-up.
Measure: Median (Inter-Quartile Range); unit: μM
Arm/Group | Active Cocoa Extract | Cocoa Extract Placebo | Active Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 992 | 925 | 966 | 951
μM | 10.3 [2.1 to 36.9] | 2.9 [0.7 to 10.2] | 5.9 [1.2 to 22.3] | 5.3 [1.2 to 19.6]

17. Other Pre Specified Outcome: Systolic and Diastolic Blood Pressure
Time Frame: 2 years
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Pulse Wave Velocity and Central Blood Pressure Indices
Description: Assessed by pulse wave analysis
Time Frame: 2 years
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Physical Performance
Description: Balance tests, grip strength, timed chair stands, walking speed
Time Frame: 2 years
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Bone Mass Density in Hip, Spine, and Total Body, and Body Composition
Description: Assessed by dual x-ray absorptiometry
Time Frame: 2 years
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Body Composition
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 years
Groups:
- Placebo Cocoa Extract: Cocoa extract placebo, 2 capsules/day
- Placebo Multivitamin: Multivitamin placebo, 1 tablet/day
- Active Cocoa Extract + Active Multivitamin: Cocoa extract: 2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin and 50 mg theobromine
  Multivitamin: Multivitamin, 1 tablet/day
- Active Cocoa Extract + Placebo Multivitamin: Cocoa extract: 2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin and 50 mg theobromine
  Multivitamin placebo: Multivitamin placebo, 1 tablet/day
- Placebo Cocoa Extract + Active Multivitamin: Multivitamin: Multivitamin, 1 tablet/day
  Cocoa extract placebo: Cocoa extract placebo, 2 capsules/day
- Placebo Cocoa Extract + Placebo Multivitamin: Cocoa extract placebo: Cocoa extract placebo, 2 capsules/day
  Multivitamin placebo: Multivitamin placebo, 1 tablet/day
Arm/Group | Active Cocoa Extract | Placebo Cocoa Extract | Active Multivitamin | Placebo Multivitamin | Active Cocoa Extract + Active Multivitamin | Active Cocoa Extract + Placebo Multivitamin | Placebo Cocoa Extract + Active Multivitamin | Placebo Cocoa Extract + Placebo Multivitamin
All-Cause Mortality (participants affected / at risk) | 353/10719 | 397/10723 | 362/10720 | 388/10722 | 175/5360 | 178/5359 | 187/5360 | 210/5363
Serious Adverse Events (participants affected / at risk) | 1378/10719 | 1372/10723 | 1388/10720 | 1362/10722 | 703/5360 | 675/5359 | 685/5360 | 687/5363
Other Adverse Events (participants affected / at risk) | 9965/10719 | 9950/10723 | 9942/10720 | 9973/10722 | 4985/5360 | 4980/5359 | 4957/5360 | 4993/5363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Cocoa Extract (N=10719) | Placebo Cocoa Extract (N=10723) | Active Multivitamin (N=10720) | Placebo Multivitamin (N=10722) | Active Cocoa Extract + Active Multivitamin (N=5360) | Active Cocoa Extract + Placebo Multivitamin (N=5359) | Placebo Cocoa Extract + Active Multivitamin (N=5360) | Placebo Cocoa Extract + Placebo Multivitamin (N=5363)
Total cardiovascular event (Vascular disorders) | 410 | 456 | 429 | 437 | 206 | 204 | 223 | 233 — This outcome was a composite of myocardial infarction, stroke, CVD death, CABG/PCI, unstable angina including hospitalization, carotid artery surgery, and peripheral artery surgery
Major cardiovascular event plus CABG/PCI (Vascular disorders) | 362 | 403 | 381 | 384 | 180 | 182 | 201 | 202 — This outcome was a composite of myocardial infarction, stroke, and CVD death. CABG/PCI, coronary artery bypass graft and percutaneous coronary intervention; CVD, cardiovascular disease.
Myocardial infarction (Vascular disorders) | 88 | 101 | 96 | 93 | 47 | 41 | 49 | 52
Stroke (Vascular disorders) | 113 | 124 | 121 | 116 | 56 | 57 | 65 | 59
Death from cardiovascular causes (Vascular disorders) | 76 | 104 | 84 | 96 | 37 | 39 | 47 | 57
Coronary revascularization procedures (Vascular disorders) | 166 | 175 | 177 | 164 | 87 | 79 | 90 | 85
Unstable angina requiring hospitalization (Vascular disorders) | 46 | 46 | 50 | 42 | 26 | 20 | 24 | 22
Carotid artery disease (Vascular disorders) | 25 | 27 | 24 | 28 | 12 | 13 | 12 | 15
Peripheral artery disease (Vascular disorders) | 17 | 19 | 16 | 20 | 7 | 10 | 9 | 10
Major cardiovascular events (Vascular disorders) | 255 | 304 | 274 | 285 | 127 | 128 | 147 | 157 — This outcome was a composite of myocardial infarction, stroke, and CVD death. CVD, cardiovascular disease.
Invasive Cancer of any type (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 550 | 503 | 518 | 535 | 283 | 267 | 235 | 268
Breast cancer (in women) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 99 | 81 | 93 | 87 | 54 | 45 | 39 | 42
Prostate cancer (in men) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 113 | 93 | 93 | 113 | 54 | 59 | 39 | 54
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 38 | 29 | 38 | 29 | 22 | 16 | 16 | 13
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 49 | 58 | 41 | 66 | 18 | 31 | 23 | 35
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 39 | 35 | 34 | 40 | 20 | 19 | 14 | 21
Death from cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 116 | 109 | 116 | 109 | 58 | 58 | 58 | 51
Gastrointestinal bleeding (Blood and lymphatic system disorders) | 507 | 507 | 544 | 470 | 272 | 235 | 272 | 235
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Cocoa Extract (N=10719) | Placebo Cocoa Extract (N=10723) | Active Multivitamin (N=10720) | Placebo Multivitamin (N=10722) | Active Cocoa Extract + Active Multivitamin (N=5360) | Active Cocoa Extract + Placebo Multivitamin (N=5359) | Placebo Cocoa Extract + Active Multivitamin (N=5360) | Placebo Cocoa Extract + Placebo Multivitamin (N=5363)
Stomach upset or pain (Gastrointestinal disorders) | 5119 | 4984 | 4943 | 5160 | 2516 | 2603 | 2427 | 2557
Nausea (Gastrointestinal disorders) | 3900 | 3756 | 3827 | 3829 | 1977 | 1923 | 1850 | 1906
Constipation (Gastrointestinal disorders) | 5077 | 5143 | 5126 | 5094 | 2564 | 2513 | 2562 | 2581
Diarrhea (Gastrointestinal disorders) | 5627 | 5639 | 5521 | 5745 | 2762 | 2865 | 2759 | 2880
Skin rash (Skin and subcutaneous tissue disorders) | 3520 | 3476 | 3425 | 3571 | 1685 | 1835 | 1740 | 1736
Skin discoloration (Skin and subcutaneous tissue disorders) | 2332 | 2361 | 2294 | 2399 | 1124 | 1208 | 1170 | 1191
Fatigue or drowsiness (General disorders) | 6268 | 6228 | 6215 | 6281 | 3142 | 3126 | 3073 | 3155
Flu-like symptoms (Infections and infestations) | 3851 | 4022 | 3962 | 3911 | 1979 | 1872 | 1983 | 2039
Dizziness (General disorders) | 4195 | 4129 | 4113 | 4211 | 2075 | 2120 | 2038 | 2091
Frequent nosebleeds (Blood and lymphatic system disorders) | 524 | 555 | 533 | 546 | 258 | 266 | 275 | 280
Easy bruising (Blood and lymphatic system disorders) | 3836 | 3864 | 3756 | 3944 | 1879 | 1957 | 1877 | 1987
Blood in urine (Blood and lymphatic system disorders) | 904 | 863 | 876 | 891 | 446 | 458 | 430 | 433
Migraine (Nervous system disorders) | 834 | 971 | 887 | 918 | 409 | 425 | 478 | 493
Other headaches (Nervous system disorders) | 4010 | 4176 | 4065 | 4121 | 2007 | 2003 | 2058 | 2118
Lightheadedness (General disorders) | 4269 | 4231 | 4206 | 4294 | 2126 | 2143 | 2080 | 2151
Unintentional Fall (General disorders) | 6067 | 6059 | 6042 | 6084 | 3048 | 3019 | 2994 | 3065

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02422745/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT02422745/SAP_001.pdf